CLINICAL TRIAL: NCT01294332
Title: Effect of Aerobic Exercise Training on Cardiorespiratory Fitness in Patients With Traumatic Brain Injury
Brief Title: Effect of Aerobic Exercise Training on Cardiorespiratory Function in Patients With Traumatic Brain Injury
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: Center for Neuroscience and Regenerative Medicine (CNRM) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 110088; 11-CC-0088
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Last update posted 2025-12-31 (Actual); Status verified 2025-12-09

CONDITIONS: Exercise; Fatigue; Physical Fitness; Traumatic Brain Injury
Keywords: Cognition; TBI; Mood; Aerobic Exercise Training; Cardiorespiratory Fitness
MeSH Terms: conditions — Motor Activity; Fatigue; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): Aerobic exercise performed for 12 weeks
  Interventions: Other: Aerobic Exercise Training

INTERVENTIONS:
Other: Aerobic Exercise Training — supervised exercise on the treadmill at target heart rate range for 12 weeks, 3 times a week for 30 minutes.

SUMMARY:
Background:

- Many people who have traumatic brain injury (TBI) have low levels of physical fitness. Low physical fitness causes severe fatigue that reduces the ability to perform routine daily activities, and may also cause increased depression, anxiety, or sadness. Aerobic exercise, such as treadmill walking or running, improves physical fitness in most people and may also decrease fatigue and improve mood. However, more information is needed to determine if exercise improves these conditions in people who have TBI.

Objectives:

- To examine the effect of an aerobic treadmill walking exercise program on physical fitness, fatigue, and mood in people with TBI.

Eligibility:

- Individuals between 21 and 45 years of age who had a nonpenetrating traumatic brain injury at least 6 months before participating; able to understand oral and written English language, give informed consent and sign a consent form; are physically inactive (including activities related to both job and recreation); and are able to stand and walk on a treadmill safely without help.

Design:

* This study requires 4 testing visits and 36 exercise visits over 14 weeks.
* The first and third testing visits will last about 4 hours and the second and final testing visits will take about 2 hours.
* Testing visits will consist of a medical history and physical examination, completion of questionnaires (about fatigue, daily physical activity, sleep quality, mood, and overall quality of life), tests of thinking and a treadmill exercise test.
* Participants will have treadmill exercise training 3 days per week for 12 weeks. Each session includes a check-in, warm-up, treadmill walking at the training heart rate, and cool-down. Thirty-two of the sessions will last for about 1 hour, and four of the sessions will include questionnaires to fill out and will last about one-and-a-half hours.
* After completing the exercise training program, participants will have a final testing visit to complete the questionnaires (about fatigue, daily physical activity, sleep quality, mood, and overall quality of life), tests of thinking and a treadmill exercise test.

DETAILED DESCRIPTION:
Objective

The broad objective of this exploratory project is to inform clinical studies and trials on the use of aerobic exercise training (AET) as an intervention for improving cardiorespiratory fitness in patients with traumatic brain injury (TBI). AET-induced adaptation of cardiorespiratory fitness and fatigue severity will be characterized, and time-course for changes in mood reactivity will be determined. We hypothesize that 1) AET will improve both cardiorespiratory fitness and fatigue severity 2) mood will at first worsen in response to AET but that mood reactivity will then decrease at some point during the intervention, and 3) AET will not impair overall cognitive performance, but that the specific cognitive performance areas of attention and concentration will improve with AET.

Study Population

Thirty-six adult subjects with a clinical diagnosis of non-penetrating TBI (mild, moderate, and severe) will be enrolled. Subjects will be recruited from NIH, affiliated hospitals/clinics, and in the community.

Design

This is a pilot study with a pre-experimental, test-intervention-retest design. Cardiorespiratory fitness, fatigue severity, cognitive performance, and changes in mood reactivity will be measured at baseline. The subjects will then participate in a 12-week treadmill exercise training intervention protocol known to improve cardiorespiratory fitness in the general population. Following the 12 weeks of AET, cardiorespiratory fitness, fatigue severity, and cognitive performance will be retested and compared to baseline. Changes in mood reactivity will be assessed monthly.

Outcome Measures

AET-induced change in cardiorespiratory fitness as measured by peak oxygen consumption (VO2) is the primary outcome measure and will be measured by pulmonary gas exchange analysis during treadmill exercise tolerance testing. A submaximal, continuous work rate test will also be used to measure the ability of the cardiorespiratory system to meet the energy demands of work over time (VO2 on-kinetics). The Fatigue Severity Scale (FSS) is the principal measurement tool for the fatigue outcome variable. FSS scores will be interpreted in relation to information from the Medical Outcomes Study 36-Item Short Form (MOS-36SF), Becks Depression Inventory (BDI), The Pittsburgh Sleep Quality Index (PSQI), International Physical Activity Questionnaire (IPAQ) and the Profile of Mood States Short Form (POMS-SF). Cognitive performance will be tested and interpreted compared to norms by the Finger Tapping Test (FTT), the Trail Making Test (TMT) and the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS). Change in mood reactivity will be measured as the difference in the POMS-SF scores before and after 30 minutes of recovery. The outcome variable for time-course related change in mood reactivity is the week of onset for significant improvement in mood reactivity.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects eligible for participation in this research study must meet the following inclusion criteria:

1. Diagnosis of non-penetrating mild, moderate, or severe TBI
2. Injury occurred at least 6 months prior to enrollment
3. Age 21-45 years
4. Physically inactive as identified by a physician.
5. Able to stand and walk on a treadmill independently and safely without assistance
6. Able to follow the study protocol
7. Fluent in English and able to provide informed consent
8. Willing and safely able to forego starting or changing an exercise program or treatments that would potentially alter cardiorespiratory capacity or ability to exercise and/or treatment for mood disorders

EXCLUSION CRITERIA:

Subjects are not eligible for participation in this research study if any of the following medical conditions that would impair aerobic capacity or the ability to engage in physical activity exist, including diseases of the cardiovascular (other than hypertension controlled by medication to below 140/90 mmHg), pulmonary, neurological, metabolic, or musculoskeletal systems such as:

1. Diagnosis or history of ischemic heart disease, including those with CABG and PTCA
2. Dilated or hypertrophic cardiomyopathy
3. Non-idiopathic cardiomyopathy
4. Uncontrolled hypertension, defined as a resting blood pressure above 140/90 mmHg
5. Diagnosis or history of right or left-sided heart failure or pulmonary hypertension
6. Diagnosis or history of restrictive or obstructive lung disease
7. Diagnosis or history of stroke
8. Type I or Type II Diabetes Mellitus
9. Diagnosis of chronic kidney disease, chronic liver disease, acute kidney injury or acute liver failure
10. Metastatic cancer active within the previous five years
11. Mitochondrial disease
12. On medications that would influence aerobic capacity, the ability to adapt to exercise training, or treadmill performance such as beta blockers or antiretroviral therapy
13. Active substance abuse including ETOH
14. Ongoing tobacco use (any use within the past six months)
15. Medical or Psychological instability such that the subject could not reasonably be expected to fulfill the study requirements
16. Pregnancy
17. BMI greater than 40 kg/m(2)

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2011-05-26 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2014-02-11 (Actual)

PRIMARY OUTCOMES:
Change in peak oxygen consumption | Pre and post
  The peak VO2 as measured by gas exchange during a cardiopulmonary exercise test to volitional exhaustion.

CONTACTS AND LOCATIONS:
Overall Officials: Leighton Chan, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chin LMK, Chan L, Drinkard B, Keyser RE. Oxygen uptake on-kinetics before and after aerobic exercise training in individuals with traumatic brain injury. Disabil Rehabil. 2019 Dec;41(24):2949-2957. doi: 10.1080/09638288.2018.1483432. Epub 2018 Jun 30. PMID 29961351
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-CC-0088.html